CLINICAL TRIAL: NCT07044076
Title: Translation and Validation of the MQOL Self-questionnaire Into French for Assessing Quality of Life in Patients With Meningiomas
Acronym: MenQOL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D25 - P003
Record Dates: First submitted 2025-06-10; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life; Meningioma
MeSH Terms: conditions — Meningioma | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life — The four questionnaires (MQOL, EQ-5D, Karnofsky, and FACT-Br) will be sent to patients online using the secure online platform Redcap.

SUMMARY:
Meningiomas, which account for about 40% of primary central nervous system tumors, have significant psychological and social impacts, even without treatment. Their effect on quality of life is often underestimated and poorly documented. There is one validated questionnaire (MQOL) but it has not yet been translated into French. The project involves two phases: first, translating and linguistically validating the MQOL into French; second, scientifically validating the questionnaire with 50 meningioma patients using established scales (EQ-5D, Karnofsky, FACT-Br) to ensure its reliability and internal consistency.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Diagnosis of intracranial meningioma confirmed by imaging or surgery

Exclusion Criteria:

* Pregnant or breastfeeding women (Article L1121-5)
* Patients deprived of liberty by judicial or administrative decision, as well as individuals undergoing psychiatric care (Article L1121-6)
* Patients not fluent in French or with poor understanding of the language
* Inability to refuse participation in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of three groups to ensure maximum heterogeneity:
  1. The study will be announced to all patients seen in consultation for meningioma at GHU Paris - Sainte-Anne (France).
  2. All patients who are members of the AMAVEA association will be notified of the study by email.
  3. Any patient referred by partner teams following a call for participation within the Neuro-Oncology Club and the Skull Base Club of the French Neurosurgery Society, recruited under the same procedure as the AMAVEA association.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-07-13 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
meningioma-specific quality-of-life questionnaire | 1 month
  The meningioma-specific quality-of-life questionnaire (MQOL) is an self-administered questionnaires and a validated tool used in practice in English, specifically applicable to patients with meningiomas, and was developed by a Canadian team (Baba A, Saha A, McCradden MD, Boparai K, Zhang S, Pirouzmand F, Edelstein K, Zadeh G, Cusimano MD. Development and validation of a patient-centered, meningioma-specific quality-of-life questionnaire. J Neurosurg. 2021 May 14;135(6):1685-1694. doi: 10.3171/2020.11.JNS201761. PMID: 33990085.)
  This project will involve applying the MQOL to a population of 50 patients and comparing it with self-administered questionnaires already validated in French practice (FACT-Br, Karnofsky, and EQ-5D).
  The purpose of all these questionnaires is to assess quality of life in patients.
  The EQ-5D and Karnofsky evaluate it in a general manner, while the FACT-Br is used in an oncological context.

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris -Psychiatrie & Neurosciences, Paris, France